CLINICAL TRIAL: NCT01212627
Title: BrUOG- Phase 1-233: A Phase I Study of Ridaforolimus With Cetuximab for Patients With Advanced Head and Neck Cancer, Non-Small Cell Lung Cancer and Colon Cancer
Brief Title: Ridaforolimus With Cetuximab: Adv Non-Small Cell Lung, Colorectal, Head & Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Determination to stop enrollment made due to funding
Sponsor: Angela Taber MD (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); Memorial Hospital of Rhode Island (Other); Roger Williams Medical Center (Other)
Responsible Party: Sponsor-Investigator, Angela Taber MD, Principle Investigator, Brown University
Organization: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-Phase 1-233
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ridaforolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ridaforolimus (Experimental): Ridaforolimus: 20mg Daily, 5 days each week, on a 28 day cycle until progression
  Interventions: Drug: Ridaforolimus

INTERVENTIONS:
Drug: Ridaforolimus — Ridaforolimus 20 Daily, 5 days each week, (Mon-Fri) on a 28 day cycle
  Other Names: deforolimus

SUMMARY:
The main purpose of this study is to evaluate the best dose, safety and side effects of ridaforolimus when given with cetuximab for patients with head and neck, lung and colon cancer that has progressed after initial therapy. A second purpose of this study is to gain preliminary information on whether the combination of ridaforolimus and cetuximab is helpful in treating patients with advanced head and neck cancer

DETAILED DESCRIPTION:
Patients with advanced NSCLC, colorectal cancer, and head and neck cancer that progressed after at least 1 prior regimen for metastatic disease were eligible. Wild-type K-ras was required in colon cancer. All patients received cetuximab 400 mg/m2 week 1 followed by 250 mg/m2/week. Four dose levels of ridaforolimus were planned: 10mg, 20mg, 30mg, and 40mg daily, 5 days each week, on a 28-day cycle.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically advanced head and neck cancer, NSCLC or colorectal cancer (wild-type KRAS) in whom there is no curable option and have progressed after at least one regimen for advanced disease. Once the final dose level has been determined, only patients with advanced lung cancer who fail at least one line of chemotherapy will be eligible to be accrued to the 13 patient expanded cohort. *** As of July 7, 2011 the final dosing level has been determined and the next cohort of patients with advanced lung cancer will be enrolled**
* Patient has measurable disease by protocol-specific RECIST criteria.
* A minimum of 4 weeks has elapsed between prior chemotherapy and day 1 of study treatment.
* A minimum of 14 days has elapsed since prior kinase inhibitor therapy or radiotherapy, and a minimum of 4 weeks has elapsed since prior bevacizumab.
* No prior exposure to an mTOR inhibitor. Prior cetuximab exposure is allowed.
* ECOG performance status 0-1
* Required initial lab values: Hemoglobin ≥9.0 g/dL, absolute neutrophil count ≥1,500/mm3, platelet count ≥100,000/mm3, total bilirubin ≤1.5 times the upper limit of normal, AST or ALT <3 times the upper limit of normal, serum albumin ≥2.5 g/dL, serum cholesterol ≤350 mg/dL, triglycerides ≤400 mg/dL, creatinine <1.5 times the upper limit of normal, or a calculated creatinine clearance ≥50 ml/min.
* Age ≥18 years
* Those of child-bearing potential must agree to use of effective method of contraception
* Patients must have the ability to understand and give written informed consent

Exclusion criteria:

* Patient is known to have active brain metastases. Patients with previously treated brain metastases that are stable for >3months are eligible if a current brain MRI (within 28 days of day 1 of study treatment) shows no edema or evidence of progression compared to a prior study at least 3 months ago.
* Patient is currently participating or has participated in a study with an investigational anticancer treatment or device within 30 days or 5 half lives of the investigational compound (whichever is greater) of initial dosing with study drug.
* Patient has previously received rapamycin or rapamycin analogs, including ridaforolimus, everolimus, or temsirolimus.
* Patient is receiving corticosteroids administered at doses greater than those used for normal replacement therapy.
* Patient has a history of prior invasive malignancy except for basal cell carcinoma of the skin within the past two years or who is deemed at low risk for recurrence by his treating physician.
* Patient has known severe hypersensitivity to macrolide antibiotics (ie: clarithromycin, erythromycin, or azythromycin).
* Patient has NYHA Class III or IV congestive heart failure or any other significant history of cardiac disease including: myocardial infarction within the last 6 months; ventricular arrhythmia or acute congestive heart failure within the last 3 months; uncontrolled angina or uncontrolled hypertension.
* Patient is known to be HIV positive or has a known history of Hepatitis B or C.
* Patient has a psychiatric disorder that would interfere with cooperation with the requirements of the trial, is a regular user of illicit drugs (including "recreational use"), or has a recent history (within the last year) of drug or alcohol dependence.
* Patient is pregnant or breastfeeding, or expecting to conceive within the projected duration of the study.
* Patient has an active infection requiring intravenous antibiotics.
* Patient has a requirement for concurrent treatment with medications that are strong inducers or inhibitors of cytochrome P450 (CYP3A) (see Appendix). Patients should discontinue these medications for at least 2 weeks prior to the first dose of ridaforolimus. Concomitant medications that are metabolized by CYP3A are allowed (e.g., simvastatin or atorvastatin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Plette, MD, Principal Investigator — Lifespan
Locations (2):
- United States (2):
  - memorial Hospital of Rhode island, Pawtucket, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Ridaforolimus,: Ridaforolimus: 20mg Daily, 5 days each week, on a 28 day cycle until progression
  Ridaforolimus: Ridaforolimus 20 Daily, 5 days each week, (Mon-Fri) on a 28 day cycle
  Ridaforolimus
Period: Overall Study
Arm/Group | Ridaforolimus,
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ridaforolimus,
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 57.8 [42 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Determine Maximum Tolerated Dose (MTD) of Ridaforolimus With Given With Cetuximab
Description: the first testing will occur once the first 3 patients are enrolled and have received 1 cycle DLT's will be evaluated- if everything is ok then the next level of medication will begin
  Weekly Ridaforolimus Dose Level 1 20 mg/day Dose Level 2 30 mg/day Dose Level 3 40 mg/day
Time Frame: 1 year
Measure: Number; unit: mg/day
Arm/Group | Ridaforolimus,
Number analyzed (Participants) | 12
mg/day | 20

2. Secondary Outcome: Check the Tolerability, and Maximum Tolerated Dose (MTD) of Several Dosing Schedules of Oral Ridaforolimus.
Description: the first testing will occur once the first 3 patients are enrolled and have received 1 cycle DLT's will be evaluated- if everything is ok then the next level of medication will begin
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline, treatment, 30 days post last dose of drug
Arm/Group | Ridaforolimus,
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ridaforolimus, (N=12)
acute renal failure (Investigations) | 1 (1)
Anemia (Investigations) | 1 (1)
aspiration (Investigations) | 1 (1)
ejection fraction (Investigations) | 1 (1)
Hypokalemia (Investigations) | 1 (1)
pericardial effusion (Investigations) | 1 (1)
Pleural Effusion (Investigations) | 1 (1)
pneumonia (Investigations) | 1 (1)
Respiratory Failure (Investigations) | 1 (1)
Shortness of Breath/dyspnea (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ridaforolimus, (N=12)
acne (Investigations) | 2 (2)
Alk phos (Investigations) | 3 (3)
Anemia (Investigations) | 10 (10)
Anorexia (Investigations) | 3 (3)
change in taste (Investigations) | 2 (2)
Constipation (Investigations) | 3 (3)
cough (Investigations) | 4 (4)
Dehydration (Investigations) | 2 (2)
despression (Investigations) | 1 (1)
Diarrhea (Investigations) | 2 (2)
Dry skin/pruritis/cracked skin (Investigations) | 8 (8)
dysphagia (Investigations) | 1 (1)
edema (Investigations) | 2 (2)
Epistaxis (Investigations) | 2 (2)
Fatigue (Investigations) | 7 (7)
Facial Hair growth (Investigations) | 1 (1)
headache (Investigations) | 2 (2)
hiccups (Investigations) | 1 (1)
Hyperbilirubinemia (Investigations) | 1 (1)
hypercholesterolemia (Investigations) | 5 (5)
hypersensitivity reaction (Investigations) | 2 (2)
hypoalbuminemia (Investigations) | 8 (8)
Hyponatremia (Investigations) | 6 (6)
hypocalcemia (Investigations) | 6 (6)
hypoglycemia (Investigations) | 3 (3)
Hypokalemia (Investigations) | 4 (4)
Hypomagnesemia (Investigations) | 6 (6)
Hypotension (Investigations) | 2 (2)
Increased phosp (Investigations) | 2 (2)
Increased PT/INR (Investigations) | 4 (4)
infection (Investigations) | 5 (5)
Ingrown nail- toe (Investigations) | 1 (1)
Lipase (Investigations) | 1 (1)
LFTs (Investigations) | 3 (3)
Lymphopenia (Investigations) | 5 (5)
Light headedness/dizzy (Investigations) | 1 (1)
Mucositis (Investigations) | 7 (7)
nail changes (Investigations) | 1 (1)
Nausea (Investigations) | 7 (7)
Neuropathy (Investigations) | 5 (5)
Pain-localized (Investigations) | 6 (6)
Pain-general (Investigations) | 1 (1)
Pain-chest (Investigations) | 1 (1)
Pink eyelid (Investigations) | 1 (1)
Pleural Effusion (Investigations) | 1 (1)
Post nasal drip (Investigations) | 1 (1)
Rash (Investigations) | 8 (8)
Shortness of Breath/dyspnea (Investigations) | 3 (3)
sore throat (Investigations) | 1 (1)
Thrombocytopenia (Investigations) | 4 (4)
TSH (Investigations) | 1 (1)
Thrush (Investigations) | 1 (1)
Triglycerides (Investigations) | 5 (5)
Vomitting (Investigations) | 2 (2)
WBC (Investigations) | 4 (4)
wt loss (Investigations) | 2 (2)
uric acid (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No